CLINICAL TRIAL: NCT06872710
Title: Prognostic Value of Vitamin D and IPTH in Pulmonary Hypertension
Brief Title: Prognostic Value of Vitamin D and Intact Parathyroid Hormone (iPTH) in Pulmonary Hypertension
Acronym: NBHAP
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Francisco Pérez Vizcaíno, Full professor, Universidad Complutense de Madrid
Other Study IDs: 14/2023; REHAP (Registry Identifier: Registro Español de Hipertensión Arterial Pulmonar); REHAR (Registry Identifier: Registro Español de Hipertensión pulmonar Asociada a enfermedad Respiratoria)
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Hypertension
Keywords: Vitamin D; iPTH; hyperparathyroidism
MeSH Terms: conditions — Hypertension, Pulmonary; Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 13 Years
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Control: 46 anonymized serum samples from controls without any known cardiovascular disease collected at the Biobank, matched by sex and age with the other cohorts. All the available samples were recruited. This group is used to compare the biomarker levels in healthy individuals.
- Pulmonary arterial hypertension (group 1 PH): 170 anonymized serum samples from patients with pulmonary arterial hypertension, including patients with idiopathic PAH (87), heritable PAH (5), drug-induced PAH (8), PH associated to connective tissue disease (27), PH associated to portal hypertension (12), associated ot congenital heart disease (31). Samples were randomly selected by the Biobank administrators with the only condition that they had not been previously analyzed by us.
- Chronic thromboembolic pulmonary hypertension (group 4 PH): 100 anonymized serum samples from patients with chronic thromboembolic pulmonary hypertension.
- Pulmonary hypertension associated to Chronic Respiratory Disease or hypoxia (group 3 PH): 30 anonymized serum samples from patients with CRD-associated PH. All the available samples were recruited.

INTERVENTIONS:
Other:  — There are no interventions. Samples were collected by the Biobank since 2013.

SUMMARY:
The aim of this observational study is to analyse the prognostic value of 25(OH)-vitamin D, iPTH and other serum biomarkers in patients with pulmonary hypertension.

Serum samples are obtained from the Spanish Biobank of pulmonary hypertension. Clinical data will be collected from the Spanish registries on pulmonary hypertension (REHAP and REHAR).

DETAILED DESCRIPTION:
Background. Pulmonary hypertension (PH) is a heterogeneous pathophysiological condition characterized by progressive pulmonary vascular narrowing that ultimately results in right-sided heart failure and eventually death or lung transplantation.

Pulmonary arterial hypertension (PAH, group 1 PH), PH associated to chronic respiratory diseases or hypoxia (CRDPH, group 3 PH) and chronic thromboembolic pulmonary hypertension (CTEPH, group 4) are subgroups of pulmonary hypertension.

The effectiveness of current pharmacological treatments is suboptimal and a large proportion of patients still had events or died despite receiving combination therapy. Vitamin D deficiency has been found to be much more frequent in PAH patients than in the general population or even compared to patients with other severe cardiovascular diseases. Our previous study (PMID: 32041235) showed that PAH deficiency has a negative prognostic impact in three subgroups of PAH (idiopathic, heritable and drug-induced). Animal studies support that vitamin D deficiency worsens PAH.

Serum samples are available from the Spanish Biobank of pulmonary hypertension in IDIBAPS (Hospital Clinic, Barcelona) which has collected and stored samples from Spanish PH patients since 2013. The samples are anonymized and linked to clinical data, which are recorded in the registries REHAP (group 1 and 4 PH) and REHAR (group 3 PH) and are continuously updated.

Biomarkers, including, but not limited, to 25-OH-vitamin D and iPTH, will be measured in the samples using commercial ELISA kits. These measured values will be related to the clinical variables. Patients will be classified according to the biomarker levels. The analysis of the Receiver operating characteristic (ROC) curve will be performed and the optimal cutoff values for biomarkers levels will be chosen based for each biomarker.

The main end-point of the study is to analyze whether the levels of a given serum biomarker predicts survival as analyzed by a Kaplan-Meier analysis and statistically compared using the log-rank test.

Secondary end-points. The Cox's proportional hazards model will be also used to include additional covariates. Additional variables that will be compared: 6-min walking distance, tricuspid annular plane systolic excursion (TAPSE), B-type natriuretic peptide (BNP) and the N-terminal fragment of pro-BNP (NT-pro-BNP) levels, New York Heart Association (NYHA) functional class, the non-invasive risk score (PMID: 28775050).

Two-sample comparisons will be analyzed using Mann-Whitney test for non normal continuous variables, t-test for normal continuous variables, and exact Fisher test or chi-square for trends for NYHA functional class or risk assessment. Data will be presented as scatter plots and medians. A p-value less than 0.05 will be considered statistically significant.

This is a collaborative study within the Ciberes Network Francisco Pérez Vizcaíno (Univ Complutense) Isabel Blanco (IDIBAPS) Rui Adao (Univ Complutense)

ELIGIBILITY:
Inclusion Criteria: Samples from patients with group 1, 3 or 4 PH stored in the Spanish PH Biobank (IdiBAPS). A maximum of 100 samples was limited for PAH associated to groups 1.1, 1.2 and 1.3 (idiopathic, heritable and drug-induced PH) and 100 samples from group 4. Samples will be randomly selected by the Biobank managers. All available samples from control (matched for sex and age) and group 3 PH.

Exclusion Criteria:

1. Samples from PAH associated to HIV infection, schistosomiasis or PAH with features of venous/capillary (PVOD/PCH) involvement.
2. Samples from patients that were analyzed in our previous study (PMID: 32041235)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed of PH (groups 1, 3 and 4) which have donated serum samples to the Spanish Biobank of PH. All these patients are included in the Spanish registries of PH (REHAP for groups 1 and 4, REHAR for group 3) Samples available in the Biobank from controls who have donated serum and have no known cardiovascular disease.
Sampling Method: Probability Sample
Enrollment: 345 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Survival | Events (deaths) will be analyzed from the blood sample extraction until March 1st 2025.
  The main end-point of the study is to analyze whether the levels of the serum biomarker predicts survival as analyzed by a Kaplan-Meier analysis and statistically compared using the log-rank test.

SECONDARY OUTCOMES:
Survival (hazard risk) and transplant-free survival | Events (death or transplant) will be analyzed from the blood sample extraction until March 1st 2025.
  Survival will also be analyzed using the Cox's proportional hazards model to analyze potential co-variates.
  To analyze whether the levels of the serum biomarker predicts transplant-free survival as analyzed by a Kaplan-Meier analysis and statistically compared using the log-rank test.
Clinical risk factors | Parameters will be obtained from the registry at the nearest date within six months of the date of plasma sampling in the Biobank
  Additional variables that will be compared: 6-min walking distance, tricuspid annular plane systolic excursion (TAPSE), B-type natriuretic peptide (BNP), the N-terminal fragment of pro-BNP (NT-pro-BNP) levels, New York Heart Association (NYHA) functional class and the non-invasive risk score (PMID: 28775050).
  Two-sample comparisons will be analyzed using Mann-Whitney test for non normal continuous variables, t-test for normal continuous variables, and exact Fisher test or chi-square for trends for NYHA functional class or risk assessment. Data will be presented as scatter plots and medians. A p-value less than 0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Perez Vizcaino, PhD, Principal Investigator — Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: No
The clinical data is available in the registries REHAP and REHAR. The access to these data requires an application.